CLINICAL TRIAL: NCT06717386
Title: Modified Diagonal Pelvic Osteotomy and External Fixator in the Surgical Treatment of Bladder Exstrophy
Brief Title: Pelvic Osteotomy in Bladder Exstrophy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ali Abdelaal Bakheet, assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-24-11-1MD
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Bladder Exstrophy
MeSH Terms: conditions — Bladder Exstrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bladder epithpidius complex (Other): diagonal pelvic osteotomy in bladder exstrophy
  Interventions: Procedure: diagonal pelvic osteotomy
- bladder exstrophy (Other): horizontal pelvic osteotomy
  Interventions: Procedure: diagonal pelvic osteotomy

INTERVENTIONS:
Procedure: diagonal pelvic osteotomy — supraacetabular pelvic osteotomy in oblique shape

SUMMARY:
The study focuses on the surgical treatment of bladder exstrophy, a congenital condition where the bladder is located outside the body. It examines the use of modified diagonal pelvic osteotomy combined with an external fixator as a treatment approach. This method aims to improve pelvic support and facilitate proper bladder reconstruction. The study likely evaluates the outcomes, complications, and overall effectiveness of this surgical technique in enhancing patient quality of life and functional results. Key findings may include insights into recovery times, rates of successful bladder closure, and potential long-term benefits for patients.

ELIGIBILITY:
Inclusion Criteria:

1. age: all cases of delayed exstrophy repaior
2. sex : both gender
3. children who received no operative treatment befor

Exclusion Criteria:

1. previous pelvic surgery
2. sever comorbidities

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-12-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
symphyseal diastaisis | 1 year
  radiological

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt